CLINICAL TRIAL: NCT06962124
Title: The Effect of Accurate Measurement of Dry Weight Based on pre_dialysis Serum Sodium Measurement on Reduction of Hemodialysis Complications
Brief Title: How to Prevent Complications During Dialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Raafat Helmy, The effect of accurate measurement of dry weight based on pre_dialysis serum sodium measurement on reduction of hemodialysis complicationsAssiut, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: complications during dialysis
Record Dates: First submitted 2025-04-21; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Dialysis Related Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of measurement of dry weight based on pre dialysis serum sodium measurment on reduction of h (Experimental): measurement of dry weight based on pre dialysis serum sodium
  Interventions: Other: serum sodium measurment

INTERVENTIONS:
Other: serum sodium measurment — serum sodium measurment

SUMMARY:
We aimed to determine the effect of accurate assessment of dry weight based on measuring blood sodium level before dialysis to evaluate the effect of adjustment of ultrafiltration rate on hemodialysis complications and take a step forward to improve patient care and the quality of hemodialysis.

DETAILED DESCRIPTION:
Dialysis has become an integral part of daily routine for kidney failure patients. so, if we can reduce complications during sessions, we will reduce the burden of life as a whole ¬. Haemodialysis problems are frequent (1).

The definitions of dry weight have changed over time but can be defined as the lowest post-dialysis weight tolerated without significant signs of hypovolaemia.(2) It should be mentioned that the incidence of complications during hemodialysate depends on the balance between the rate of ultrafiltration and changes in plasma volume. The amount of ultrafiltration is typically determined by calculating the patient's dry weight.(3) Common problems during haemodialysis, in order of frequency, are: hypotension of around 23%, muscle cramps of roughly 10 to 20%, and nausea and vomiting of 10%. (4, 5). About 60 to 90% of dialysis patients suffer fatigue, which is one of the most prevalent complaints in people receiving hemodialysis.(6) aggressive ultrafiltration and targeting an inappropriately low dry weight can lead to intradialytic hypotension (IDH), nausea, central nervous system dysfunction, cramping, and risks compromising vascular access and worsening residual renal function.(7) Determining the patients' accurate dry weight is essential to minimizing these issues. When dry weight is accurately determined, quick variations in blood volume are avoided, which lowers the risk of problems during haemodialysis(8). The measurement of arterial natriuretic peptide (half-life of approximately 2 to 4 minutes), cyclic guanidine monophosphate, the diameter of the inferior vena cava (by echocardiography), bioimpedance (based on resistance measurement), and blood volume (by tracking changes in serum protein and hemoglobin) are used to determine dry weight.(9, 10) These techniques frequently need specialized equipment and are expensive. However, one practical way to measure dry weight prior to dialysis is to measure the amount of sodium, the most prevalent cation in extracellular fluid .(11)

ELIGIBILITY:
Inclusion Criteria:

- 6- not dependent to mechanical ventilation

1. at least one year history of hemodialysis
2. adults aged 18 to 65 years old
3. ability to communicate verbally
4. with no history of diabetes mellitus, urinary incontinence syndrome, heart and liver failure, and adrenal hypertrophy 5 -no use of antihypertensive and antispasmodic drugs four hours before dialysis

Exclusion Criteria:

1- Impaired consciousness 2- participant's withdrawal from the study 5-death 3- severe blood supply problem in the fistula or vascular access 4-migration or travel during the study

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
predict correlation between accurate measurement of dry weight in kilogram by predialytic serum sodium level and incidence of complications. | 3 month ( 39 session for each patient , 13 session per month)
  We aimed to determine the effect of assessment of dry weight based on measuring blood sodium level before dialysis to evaluate the effect of adjustment of ultrafilteration rate on haemodialysis complications and take a step forward to improve patient care and the quality of hemodialysis

IPD SHARING:
Plan to Share IPD: No